CLINICAL TRIAL: NCT02937038
Title: Reference Values and Determinants of Hydration in Children 3-13 y
Acronym: HYBISKUS
Status: Terminated | Type: Observational
Why Stopped: COVID-19 difficulties recruiting
Sponsor: Arizona State University (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Principal Investigator, Stavros Kavouras, Professor of Nutrition, Arizona State University
Other Study IDs: 16-02-574
Record Dates: First submitted 2016-10-12; First posted 2016-10-18 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Dehydration
Keywords: Urine Biomarkers; Child Nutrition; Hydration; Parent Nutrition Habits
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Kids 3-13 y: Healthy boys and girls of 3-13 y of age
- Parents 20-50 y: One of their Parents 20-50 y of age

SUMMARY:
Purpose:

1. Develop reference values for hydration biomarkers for children of 3 to 13 years old
2. Explore the association between children's and parents' hydration markers and fluid intake habits in children aged 3-13 y
3. Evaluate the equivalence of spot urine osmolality to 24h urine osmolality in children aged 3-13 y
4. Evaluate the differences in hydration markers between school and non-school days in children aged 3-13 y
5. Examine the role of different foods and fluids on hydration in children (3-13 y) and parents

DETAILED DESCRIPTION:
Recent studies in children have indicated that greater water intake and/or lower urine concentration are associated with better overall nutrition, increased physical activity, improved mood state, and enhanced cognition; which is specifically related to superior attention and memory when compared to sub-optimally hydrated children. Separately, ancillary water is being investigated as a potential treatment possibility for pediatric obesity. Although, causality cannot be directly confirmed, it is apparent that ample water intake in children, above and beyond the body's compensatory mechanisms, is preferable for psychological and physiological health. However, the prevalence of failure to meet water recommendations and hypohydration in children remains high. Still it is unclear if elevated hypohydration reports within the pediatric population are due to a general failure of children to meet water recommendations, or due to inadequacy of the published guidelines

ELIGIBILITY:
INCLUSION CRITERIA:

* Boys and girls aged 3-13 years old
* Parent willing to participate as a subject as well
* Parents: aged 20-50
* Children and parents willing to collect urine samples and store them at room temperature
* Avoid strenuous exercise on day of collection
* Parent: included if >50% of grocery shopping, food preparation, and feeding is handled by this parent

EXCLUSION CRITERIA:

Parents & Children:

* Evidence of clinically relevant metabolic, cardiovascular, hematologic, hepatic, gastrointestinal, renal, pulmonary, endocrine or psychiatric history of disease, based on the medical history questionnaire
* Use of medication that interferes with water metabolism
* Surgical operation on digestive tract (e.g. bariatric surgery), except possible appendectomy
* Regular drug treatment within 15 days prior to start of the study
* Not willing to refrain from exercise on the day before and during urine collection
* Unwilling to collect urine
* Inability to participate in the entire study
* Pregnancy for females

Children:

* Use of Diapers
* Enuresis or use of nappies during the day or during the night

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children (3-13 y) and their Parents (20-50 y)
Sampling Method: Non-Probability Sample
Enrollment: 1454 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Urine Hydration Biomarkers | May 2019
  24 h urine osmolality (mmol/kg water) for children (3-13 y) and one of their parents's

SECONDARY OUTCOMES:
Physical Activity | May 2019
  Physical activity levels assessed by the International Physical Activity Questionnaire for both kids and parents, expressed as MET-min/week
Anthropometric Assessment | May 2019
  Body mass index (kg/m2)
Socioeconomic Assessment | May 2019
  Family information for:
  Income ($) Ethnicity Education Employment status
Water intake | May 2019
  Dietary water intake (L)
Energy intake | May 2019
  Caloric Intake (kcal)

CONTACTS AND LOCATIONS:
Overall Officials: Stavros A Kavouras, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual report for nutrition and hydration information will be provided to the volunteers